CLINICAL TRIAL: NCT06697210
Title: Efficacy of Biofilm Removal of Different Interproximal Oral Hygiene Devices Around Posterior Single Implants. A Randomized Clinical Trial
Brief Title: Oral Hygiene Tools for Biofilm Removal Around Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Andres Pascual La Rocca, DDS , PhD, Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PER-ECL-2019-01
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Hygiene; Biofilm Removal
Keywords: dental implants; interproximal hygiene; dental superfloss; oral irrigator; interproximal brushes; plaque reduction; biofilm
MeSH Terms: interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- • Dental Floss (Vitis®, Dentaid, Barcelona, Spain). (Active Comparator): dental floss is used as interproximal hygiene device. The intervention includes thorough instruction on the correct flossing technique around dental implants to ensure effective removal of plaque and debris. Participants will be supplied with dental floss and given detailed guidance on integrating flossing into their daily oral hygiene regimen. The effectiveness of this method will be evaluated by measuring plaque levels before and after the intervention.
  Interventions: Device: • Dental Floss (Vitis®, Dentaid, Barcelona, Spain).
- • Superfloss (Oral B®, Procter & Gamble, USA) (Active Comparator): superfloss is used as the primary interproximal hygiene device. Superfloss is designed to clean around dental implants, bridges, and wide spaces between teeth. Participants will receive instructions on how to effectively use superfloss, which includes its unique combination of foam, regular floss, and spongy material to remove plaque and debris. The intervention will focus on demonstrating the proper technique to ensure optimal cleaning. The effectiveness of this method will be evaluated by comparing plaque levels before and after the intervention.
  Interventions: Device: • Superfloss (Oral B®, Procter & Gamble, USA)
- • Oral irrigator (Waterpick®, Water Pik, Inc., CO., USA) (Active Comparator): oral irrigator used as the primary interproximal hygiene device. The oral irrigator delivers a stream of pulsating water to help remove plaque and food particles from around dental implants and between teeth. Participants will receive guidance on how to properly use the oral irrigator, including the appropriate pressure settings and angles for effective cleaning. The intervention aims to enhance oral hygiene by providing a thorough rinse of the interproximal areas. The effectiveness of this method will be assessed by comparing plaque levels before and after the intervention.
  Interventions: Device: • Oral irrigator (Waterpick®, Water Pik, Inc., CO., USA)
- • Interproximal brushes (Interprox®, Vitis, Dentaid, Spain) (Active Comparator): interproximal brush is used as the primary interproximal hygiene device. The interproximal brush is specifically designed to clean between teeth and around dental implants, effectively removing plaque and debris in areas that traditional toothbrushes may miss. Participants will receive instructions on how to select the appropriate brush size and how to use it effectively to ensure optimal cleaning. The intervention will emphasize the importance of thorough brushing technique for maintaining oral health. The effectiveness of this method will be evaluated by comparing plaque levels before and after the intervention.
  Interventions: Device: • Interproximal brushes (Interprox®, Vitis, Dentaid, Spain)

INTERVENTIONS:
Device: • Dental Floss (Vitis®, Dentaid, Barcelona, Spain). — Dental Floss: A piece of dental floss approximately 40-50 cm in length was taken and placed between the index and middle fingers of each hand, leaving about 2-3 cm free in the middle. The floss was then inserted, embracing the mesial and distal surfaces, and moved up and down three times on each side
  Arms: • Dental Floss (Vitis®, Dentaid, Barcelona, Spain).
Device: • Superfloss (Oral B®, Procter & Gamble, USA) — Superfloss: The stiffened end was used to introduce the thread and the spongy-floss into the interproximal area on both the mesial and distal parts, and a gentle back-and-forth motion was applied to remove bacterial plaque. The spongy-floss was then pulled through to the regular floss section and gently slid under the gumline, followed by an up-and-down motion. These movements were repeated three times on each side.
  Arms: • Superfloss (Oral B®, Procter & Gamble, USA)
Device: • Oral irrigator (Waterpick®, Water Pik, Inc., CO., USA) — Oral Irrigator: The finest tip was selected and placed in the mesiobuccal, distobuccal, mesiolingual, and distolingual interproximal spaces. The irrigator was activated at medium power (2/3), and the process was repeated three times on each side for five seconds.
  Arms: • Oral irrigator (Waterpick®, Water Pik, Inc., CO., USA)
Device: • Interproximal brushes (Interprox®, Vitis, Dentaid, Spain) — Interproximal Brush Group: According to the interproximal space, the appropriate size was selected for each case. The brush was then placed horizontally in the interproximal space mesially and distally, and a back-and-forth movement was performed three times on each side.
  Arms: • Interproximal brushes (Interprox®, Vitis, Dentaid, Spain)

SUMMARY:
The objective of this clinical trial is to determine which interproximal hygiene device is most effective at eliminating dental plaque on implants. The main questions to be answered are:

Which interproximal hygiene device is most effective in reducing dental plaque (dental floss, superfloss, irrigator, or interproximal brush)? The researchers will compare the different devices using a plaque disclosing agent and standardized photography.

Participants:

Participants will attend a visit where the screw-retained crown will be removed, and the subgingival area will be stained with a plaque disclosing agent. The first photograph will be taken, and then the crown will be replaced. Subsequently, one of the four methods will be used randomly. The crown will be removed again, and a second photograph will be taken.

DETAILED DESCRIPTION:
The present investigation was designed as a randomized clinical trial and approved by the Ethics Committee of the Universitat Internacional de Catalunya (Barcelona, Spain) (Protocol reference PER-ECL-2019-01). The study was performed in accordance with the Declaration of Helsinki for research involving humans. After being informed about the study procedures, all patients read and signed an appropriate informed consent document prior to being included. The CONSORT guidelines for randomized clinical trials were followed.

Participants:

Periodontally healthy patients with at least one single screw-retained implant-supported crown (loaded for more than one year) on a molar or premolar site with neighboring teeth were recruited. The implants had to present ≤ 4 mm of probing pocket depth and have an appropriate prosthetic design allowing proper oral hygiene. Subjects were excluded under the following conditions: (1) drug consumption that could cause gingival enlargement, such as phenytoin, cyclosporin, and/or calcium channel blockers; (2) presence of uncontrolled diabetes mellitus; (3) smokers; (4) presence or signs of peri-implant diseases or uncontrolled periodontal disease; and (5) prosthetic design that did not allow for proper interproximal hygiene (determined by using the smallest size of interproximal brush).

One calibrated investigator (C.T.) consecutively evaluated patients for screening and was responsible for enrollment. The clinician conducted an anamnesis of the patient's medical history and recorded the clinical information.

Subsequently, patients were randomly assigned to one of the following treatment groups:

Dental Floss (Vitis®, Dentaid, Barcelona, Spain) Superfloss (Oral B®, Procter & Gamble, USA) Oral Irrigator (Waterpick®, Water Pik, Inc., CO., USA) Interproximal Brushes (Interprox®, Vitis, Dentaid, Spain) Randomization was performed using a computer-generated randomization list with permuted blocks of four, and the allocation was concealed using opaque envelopes labeled with the patient study number, which were opened just before the commencement of the intervention.

During the visit, the full mouth plaque index (FMPI) and modified plaque index at the implant site (mPI) were recorded (Mombelli et al., 1987). The mPI was assessed as follows:

Score 0: No detection of plaque. Score 1: Plaque only recognized by running a probe across the smooth marginal surface of the implant.

Score 2: Plaque visible to the naked eye. Score 3: Abundance of soft matter.

A line was drawn on the implant-supported crown with a permanent marker following the outline of the gingival margin to delimit the supragingival from the subgingival part of the crown. The screw-retained implant-supported prosthesis was subsequently removed with caution to avoid touching the interproximal areas and the cervical third of the crown, and an individualized silicone key for fixing and positioning the crown was made. Erythrosine was applied to the cervical third of the prosthesis, washed with a water syringe, and replaced in the silicone key. A standardized picture (Canon EOS 750D with annular flash Yongnuo YN14EX and macro Canon lens EF 100mm 1:28 at a distance of 44 cm and macro at 3 1.60 0.49) of the apical/subgingival third of the prosthesis was taken (Pre-area). This picture was acquired so that the plane containing the prosthetic margin was parallel to the ground and to the focal plane of the camera. The prosthesis was then replaced and screwed. At this point, the prosthesis was cleaned by the instructed operator (CT) using one of the four devices as follows:

Dental Floss: A piece of about 40-50 cm of dental floss was taken and placed between the index and middle fingers of each hand, leaving about 2-3 cm free in the middle. The dental floss was inserted, embracing the mesial and distal surfaces, and flossing up and down three times on each side.

Superfloss: The stiffened end was used to introduce the thread and the spongy-floss between the interproximal areas in both the mesial and distal parts, and a soft back-and-forth motion was applied to remove bacterial plaque. The spongy-floss was then pulled through to the regular floss section, slid gently under the gumline, and followed by an up-and-down motion. These movements were repeated three times on each side.

Oral Irrigator: The finest tip was selected and placed in the mesiobuccal, distobuccal, mesiolingual, and distolingual interproximal spaces. The irrigator was activated at medium power (2/3), and the process was repeated three times on each side for five seconds.

Interproximal Brush: According to the interproximal space, the appropriate size was selected for each case. The brush was placed horizontally in the interproximal space mesially and distally, and a back-and-forth movement was performed three times on each side.

After the interproximal cleaning was completed, the crown was unscrewed again, and a second standardized photograph was taken after removal of the crown and replaced using the silicone key with the same parameters as before (Post-area).

Image Analysis The examination was conducted based on two standardized photographs. The first photograph refers to the erythrosine-stained area of biofilm on the prosthesis at the time of removal before performing the interproximal cleaning. The second photograph refers to the residual erythrosine-stained area of the biofilm on the prosthesis at the time of removal after interproximal hygiene. Image analysis was performed using Image J® software (image processing analysis). In the first photograph, the total area delimited by the drawn margin was calculated. Subsequently, the erythrosine-colored area was delimited, determining the biofilm percentage (Pre-area). In the second picture, the residual stained area (Post-area) was calculated in the same way. The percentage reduction of plaque between the two images was then calculated.

An experienced professional (C.T.) performed the image analysis. A calibration exercise was conducted by repeating the area assessment with 40 samples, resulting in high inter-examiner reproducibility (Cronbach's α = 0.98).

Statistical Analysis Qualitative variables were described with absolute frequencies and percentages. The description of quantitative variables was performed using the mean and standard deviation (SD). The Kolmogorov-Smirnov test was used to assess the normality of distributions. Patient characteristics and clinical variables were compared according to the study groups. For the qualitative variables, the chi-squared test (Fisher exact test correction in the event of expected frequencies < 5) was used. The ANOVA test was performed to compare quantitative variables (Kruskal-Wallis test for variables with a non-normal distribution). The Bonferroni test for multiple comparisons was also performed. The intragroup biofilm reduction was analyzed using the Wilcoxon test and was also compared according to the variables of interest using the T-Student test (or U-Mann Whitney test).

The analyses were performed using R Studio software (V2.5.1). For all tests, a statistically significant difference was set at P < .05.

ELIGIBILITY:
Inclusion Criteria:

Periodontally healthy patients with at least one single screw-retained implant-supported crown (loaded for more than one year) on a molar or premolar site with neighboring teeth were recruited. The implants had to present ≤ 4 mm of probing pocket depth and have an appropriate prosthetic design that allowed for proper oral hygiene.

Exclusion Criteria:

Drug consumption that could cause gingival enlargement, such as phenytoin, cyclosporin, and/or calcium channel blockers.

Presence of uncontrolled diabetes mellitus. Smokers. Presence or signs of peri-implant diseases or uncontrolled periodontal disease. Prosthetic design that did not allow for proper interproximal hygiene (determined by using the smallest size of interproximal brush).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Biofilm reduction | Immediate Post-Treatment Evaluation: Directly after the treatment is completed to assess immediate effects.
  In the first photograph, the total area within the drawn margin was calculated.Subsequently, the erythrosine-coloured area was delimited, determining the biofilm percentage (Pre-area). In the second picture, the residual stained area (Post-area) was calculated in the same way. The percentage reduction of plaque between the two images was then calculated

CONTACTS AND LOCATIONS:
Overall Officials: Andres Pascual La Rocca, PhD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Currently under evaluation of the potential for sharing IPD and will make a decision based on ethical considerations and data protection regulations.

REFERENCES:
- [Background] Slot DE, Valkenburg C, Van der Weijden GAF. Mechanical plaque removal of periodontal maintenance patients: A systematic review and network meta-analysis. J Clin Periodontol. 2020 Jul;47 Suppl 22:107-124. doi: 10.1111/jcpe.13275. PMID 32716118
- [Background] Sirinirund B, Siqueira R, Li J, Mendonca G, Zalucha J, Wang HL. Effects of crown contour on artificial biofilm removal efficacy with interdental cleaning aids: An in vitro study. Clin Oral Implants Res. 2023 Aug;34(8):783-792. doi: 10.1111/clr.14105. Epub 2023 Jun 3. PMID 37269176
- [Background] Worthington HV, MacDonald L, Poklepovic Pericic T, Sambunjak D, Johnson TM, Imai P, Clarkson JE. Home use of interdental cleaning devices, in addition to toothbrushing, for preventing and controlling periodontal diseases and dental caries. Cochrane Database Syst Rev. 2019 Apr 10;4(4):CD012018. doi: 10.1002/14651858.CD012018.pub2. PMID 30968949
- [Background] Pons R, Nart J, Valles C, Salvi GE, Monje A. Self-administered proximal implant-supported hygiene measures and the association to peri-implant conditions. J Periodontol. 2021 Mar;92(3):389-399. doi: 10.1002/JPER.20-0193. Epub 2020 Aug 18. PMID 32761897
- [Result] van Velzen FJ, Lang NP, Schulten EA, Ten Bruggenkate CM. Dental floss as a possible risk for the development of peri-implant disease: an observational study of 10 cases. Clin Oral Implants Res. 2016 May;27(5):618-21. doi: 10.1111/clr.12650. Epub 2015 Aug 11. PMID 26261052